CLINICAL TRIAL: NCT00624325
Title: Subcutaneous Continuous Infusion of Interferon Alfa-2b and Ribavirin in Hepatitis C Genotype 1 Nonresponders
Acronym: SCIN-C
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Foundation for Liver Research (Other)
Responsible Party: R.J. de Knegt, Erasmus Medical Center Rotterdam
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCV 06-01; eudract 2006-000592-15
Record Dates: First submitted 2008-01-07; First posted 2008-02-27 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Chronic Hepatitis C
Keywords: genotype 1 nonresponders
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 12 MU interferon alfa-2b daily continuously subcutaneous in combination with 15 mg/kg/day ribavirin
  Interventions: Drug: interferon alfa-2b
- 2 (Experimental): 9 MU interferon alfa-2b daily continuously subcutaneous in combination with 15 mg/kg/day ribavirin
  Interventions: Drug: interferon alfa-2b
- 3 (Experimental): 6 MU interferon alfa-2b daily continuously subcutaneous in combination with 15 mg/kg/day ribavirin
  Interventions: Drug: interferon alfa-2b

INTERVENTIONS:
Drug: interferon alfa-2b — 12 MU daily continuously subcutaneous
  Other Names: Intron A
  Arms: 1
Drug: interferon alfa-2b — 9 MU daily continuously subcutaneous
  Other Names: Intron A
  Arms: 2
Drug: interferon alfa-2b — 6 MU daily continuously subcutaneous
  Other Names: Intron A
  Arms: 3

SUMMARY:
For chronic hepatitis C patients unresponsive to previous (PEG-)IFN/RBV combination therapy we propose continuous subcutaneous administration of high-dose IFN-a2b (Intron A®) for 48 weeks in combination with 15 mg/kg/day RBV (Rebetol®) and optimal management of side effects in order to maintain the highest possible dosages of both IFN-a2b and RBV for 48 weeks. We expect improved tolerability with continuous subcutaneous pump delivery of IFN-a2b compared to thrice weekly or daily subcutaneous injection of IFN-a2b, and increased antiviral activity and biologic potency due to sustained and higher levels of a fully potent interferon protein.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C genotype 1 unresponsive to (peg)interferon /ribavirin therapy
* In the past, peginterferon or conventional interferon plus ribavirin combination therapy for at least 12 weeks and less than 2-log HCV RNA decrease at week 12, HCV RNA positivity at week 24, breakthrough during therapy or relapse after therapy
* At least 12 weeks between end of (peg)interferon/ribavirin therapy and start of high-dose IFN/ribavirin therapy
* Persistent indication for antiviral therapy such as persistently elevated serum ALT or histological evidence of continuing or progressive fibrosis
* Age 18-60 years

Exclusion Criteria:

* Signs of progressive liver disease since end of previous therapy, beyond generally accepted criteria for HCV antiviral therapy:

  * serum bilirubin >35 μmol/l, albumin <36 g/l, prothrombin time >4 sec prolonged or platelets <100,000/mm3
  * decompensated cirrhosis (defined as jaundice in the presence of cirrhosis, ascites, gastric bleeding, esophageal varices or encephalopathy)
* Hepatic imaging (US, CT or MRI) with the evidence of hepatocellular carcinoma (hepatic imaging should be performed within 3 months prior to screening) or an alpha fetoprotein >50 ng/ml
* Other acquired or inherited causes of liver disease that could explain liver disease activity
* Co-infection with hepatitis B virus or human immunodeficiency virus (HIV)
* Other significant medical illness that might interfere with this study: significant cardiovascular, pulmonary or renal dysfunction, malignancy other than skin basocellular carcinoma in previous 5 years, immunodeficiency syndromes (e.g.: HIV positivity, steroid therapy, organ transplants other than cornea and hair transplant)
* History of a severe seizure disorder or current anticonvulsant use
* History of thyroid disease poorly controlled on prescribed medications
* Contra-indications for IFN and/or ribavirin:

  * Severe psychiatric disorder, such as major psychoses, suicidal ideation, suicidal attempt and/or manifest depression during previous (peg)interferon therapy. Severe depression would include the following: (a) subjects who have been hospitalized for depression, (b) subjects who have received electroconvulsive therapy for depression, or (c) subjects whose depression has resulted in a prolonged absence of work and/or significant disruption of daily functions. Subjects with a history of mild depression may be considered for entry into the protocol provided that a pretreatment assessment of the subject's mental status supports that the subject is clinically stable and that there is ongoing evaluation of the patient's mental status during the study
  * Reactivation of immunological disorders during previous therapy
  * Visual symptoms related to retinal abnormalities
  * Pregnancy, breast-feeding or inadequate contraception
  * Thalassemia, spherocytosis
* Substance abuse, such as alcohol (³80 gm/day) and I.V. drugs. If the subject has a history of substance abuse, to be considered for inclusion into the protocol, the subject must have abstained from using the abused substance for at least 2 years
* Any other condition which in the opinion of the investigator would make the patient unsuitable for enrollment, or could interfere with the patient participating in and completing the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of high-dose continuous subcutaneous infused IFN-a2b (serious adverse events, grade 4 NCI toxicity, percentage of patients completing treatment or reasons for dose adjustments). | 48 weeks

SECONDARY OUTCOMES:
HCV RNA negativity at week 48 and 24 weeks after end of treatment | 48 weeks
Biological activity of IFN-a2b | 48 weeks
Pharmacokinetics by IFN-a2b levels | 48 weeks
HCV-specific immune responses | 48 weeks
Quality of life assessment using SF-36 and SCL-90 questionnaires | 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: R.J. de Knegt, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands